CLINICAL TRIAL: NCT02064296
Title: Neuroimaging Approaches to Deconstructing Acupuncture for Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Harris, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: AcuAfference; R01AT007550 (NIH)
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia Chronic Pain
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Controls (No Intervention): Healthy pain free controls will be recruited for comparison with fibromyalgia patients.
- Non-Traditional Acupuncture (Active Comparator): 40 fibromyalgia patients will be randomized to non-traditional laser acupuncture (Vita Laser 650, Lhasa OMS). They will receive 2 treatments per week for 4 weeks.
  Interventions: Device: Laser acupuncture (Non-traditional Acupuncture)
- Traditional Acupuncture (Active Comparator): 40 fibromyalgia patients will be randomized to receive electro acupuncture (AS Super 4 digital needle stimulator, Harmony Medical Co) . They will receive 2 treatments per week for 4 weeks.
  Interventions: Device: Needle acupuncture (Traditional Acupuncture)

INTERVENTIONS:
Device: Needle acupuncture (Traditional Acupuncture) — This group will receive needle acupuncture at 3 pairs of sites. The needles will be stimulated with low intensity, low frequency electric current using a constant-current electro-acupuncture device (AS Super 4 digital needle stimulator).
  Arms: Traditional Acupuncture
Device: Laser acupuncture (Non-traditional Acupuncture) — For non-traditional acupuncture, a laser acupuncture device (Vita Laser 650, Lhasa OMS) will be positioned over all of the same acupoints used in EA. There will be no palpation prior to positioning these devices, and there will be no physical contact between device and skin.
  Arms: Non-Traditional Acupuncture

SUMMARY:
The aim of this study is to evaluate the impact of electro-acupuncture in pain processing on patients with fibromyalgia (FM). The investigators hypothesize that electro-acupuncture is effective for FM because it functions as a desensitization therapy, which when applied repeatedly over multiple treatment sessions, gradually habituates the nervous system to continuing pain and sensory signaling.

DETAILED DESCRIPTION:
This study design has two components: 1) a cross sectional assessment of brain chemistry, connectivity and response to pain in healthy controls and age- and sex-matched fibromyalgia patients, and 2) a longitudinal assessment of the same outcomes in fibromyalgia patients randomized to either electro-acupuncture (EA) or laser acupuncture.

The investigators will evaluate 80 fibromyalgia patients who will receive acupuncture treatment twice a week for 4 weeks, for a total of 8 treatments. Baseline data from these patients will be compared to results from 40 pain-free controls.

Participants will undergo experimental pain assessments as well as brain neuroimaging.

Note added after completion of study data gathering: Within the registration in ClinicalTrials.gov and the informed consent, one arm was referred to as "non-traditional acupuncture". In fact, this was a control arm, receiving mock laser acupuncture (Vita Laser 650, Lhasa OMS). They received 2 treatments per week for 4 weeks. As consented, they were told, with IRB permission, that they were receiving non-traditional laser acupuncture. This deception was essential to maintaining scientific integrity of the masking.

The laser acupuncture device (Vita Laser 650, Lhasa OMS) was positioned over all of the same acupoints used in electro-acupuncture (EA), but was turned off during treatment sessions. There was no palpation prior to positioning these devices, and there was no physical contact between device and skin.

ELIGIBILITY:
Inclusion Criteria for Fibromyalgia Participants

* Have self-reported FM symptoms for at least one year and also meet the Wolfe et al 2011 criteria for Fibromyalgia.
* Continued presence of pain more than 50% of days.
* Pain greater than a certain threshold on the Visual Analog Scale (VAS) for pain; 7-day recall; [Note: The VAS is widely used in clinical pain research and as such we chose to use it for inclusion criteria and for clinical pain assessment below. Within our group numerical ratings scales 0-100 are more commonly used in quantitative sensory assessment, and as such we chose to use NRS scales for evoked pain assessments below.]
* Willing to limit the introduction of any new medications or treatment modalities for control of FM symptoms during the study.
* Able to travel to the study site to receive acupuncture treatments up to two times weekly.
* Over 18 and under 65 years of age.
* Right-handed.
* Female.
* Capable of giving written informed consent.

Inclusion Criteria for Healthy Control Participants

* Over 18 and under 65 years of age.
* Female.
* Right-handed.
* Do not have fibromyalgia or an associated pain disorder, including: migraine, temporomandibular joint disorder (TMJ), chronic pelvic pain (CPP), or chronic fatigue syndrome (CFS).
* Pain less than a certain threshold on the Visual Analog Scale (VAS) for pain; 7-day recall
* Willing to complete all study procedures.
* Capable of giving written informed consent.

Exclusion Criteria for Fibromyalgia Participants:

* Acupuncture within last 6-months.
* Presence of a known coagulation abnormality, thrombocytopenia, or bleeding diathesis that may preclude the safe use of acupuncture.
* Presence of a concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc., or any other chronic pain condition with pain greater than fibromyalgia pain.
* Peripheral neuropathy of know cause that interferes with activities of daily living.
* History of vascular surgery in lower limbs or current lower limb vascular dysfunction.
* History of head injury with substantial loss of consciousness.
* Routine daily use of narcotic analgesics, marijuana or have a history of substance abuse in the past 24 months as determine by subject self-report.
* Stimulant medications, such as those used to treat ADD/ADHD (e.g., amphetamine/ dextroamphetamine [Adderall®], methylphenidate, dextroamphetamine), or the fatigue associated with sleep apnea or shift work (e.g., modafinil), are excluded.
* Concurrent participation in other therapeutic trials.
* Pregnant or nursing.
* Severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation, substance abuse within two years).
* Contraindications to fcMRI, fMRI, or 1H-MRS methods. These may include but are not limited to: surgical clips, surgical staples, metal implants, and certain metallic dental material. [Note: a more formal description of contraindications for MRI is present in our DSM Plan].
* Use of over the counter pain medications (NSAIDs, etc.) on the day of MRI scan.
* Use of as needed narcotic pain medication 48 hours prior to MRI scan.
* Current, habitual, or previous use within the last 12 months of artificial nails, nail enhancements, or nail extensions that cover any portion of either thumbnail. Exceptions, including brief and/or occasional use, may be permissible at the discretion of the principle investigator.
* Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator that would prevent satisfactory completion of the study protocol.
* Contraindications to the Electrostimulator device: Participants with electrical implants (i.e. pacemakers, defibrillators), cardiac rhythmic disorders, seizure disorders, any skin disorder in the vicinity of the electrode or an malignant diseases in the region of application. (Fibromyalgia participants only)

Exclusion Criteria for Healthy Control Participants:

* Have a diagnosis of fibromyalgia or meet the Wolfe et al 2011 criteria for Fibromyalgia.
* Presence of a concurrent autoimmune or inflammatory disease such as rheumatoid arthritis, systemic lupus erythematosus, inflammatory bowel disease, etc. that causes pain.
* Routine daily use of narcotic analgesics, marijuana or have a history of substance abuse in the past 24 months as determine by subject self-report.
* Stimulant medications, such as those used to treat ADD/ADHD (e.g., amphetamine/ dextroamphetamine [Adderall®], methylphenidate, dextroamphetamine), or the fatigue associated with sleep apnea or shift work (e.g., modafinil), are excluded.
* Concurrent participation in other therapeutic trials.
* Pregnant or nursing.
* Peripheral neuropathy of know cause that interferes with activities of daily living.
* History of vascular surgery in lower limbs or current lower limb vascular dysfunction.
* History of head injury with substantial loss of consciousness.
* Severe psychiatric illnesses (current schizophrenia, major depression with suicidal ideation, substance abuse within two years).
* Contraindications to fcMRI, fMRI, or 1H-MRS methods. (see above section)
* Use of over the counter pain medications (NSAIDs, etc.) on the day of MRI scan.
* Use of as needed narcotic pain medication 48 hours prior to MRI scan.
* Current, habitual, or previous use within the last 12 months of artificial nails, nail enhancements, or nail extensions that cover any portion of either thumbnail. Exceptions, including brief and/or occasional use, may be permissible at the discretion of the principle investigator.
* Any impairment, activity or situation that in the judgment of the Study Coordinator or Principal Investigator that would prevent satisfactory completion of the study protocol.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2014-12; Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E Harris, PhD, Principal Investigator — University of Michigan; Viataly Napadow, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Chronic Pain and Fatigue Research Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Murphy AE, Buchtel H, Mawla I, Ichesco E, Larkin T, Harte SE, Zhan E, Napadow V, Harris RE. Temporal Summation but Not Expectations of Pain Relief Predict Response to Acupuncture Treatment in Fibromyalgia. J Pain. 2024 Oct;25(10):104622. doi: 10.1016/j.jpain.2024.104622. Epub 2024 Jul 8. PMID 38986891

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 FM Participants were consented and eligible for the study but withdrew prior to being randomized to treatment.
Groups:
- Controls: Healthy pain free controls were recruited for comparison with fibromyalgia patients.
- Mock Laser Acupuncture: 39 fibromyalgia (FM) patients were randomized to control mock laser acupuncture (Vita Laser 650, Lhasa OMS). They received 2 treatments per week for 4 weeks. As consented, they were told, with IRB permission, that they were receiving laser acupuncture. This deception was essential to maintaining scientific integrity of the masking.
  Laser acupuncture (Non-traditional Acupuncture): For non-traditional acupuncture, a laser acupuncture device (Vita Laser 650, Lhasa OMS) was positioned over all of the same acupoints used in electro-acupuncture (EA), but was turned off during treatment sessions. There was no palpation prior to positioning these devices, and there was no physical contact between device and skin.
- Electro-Acupuncture: 40 fibromyalgia patients were randomized to receive electro-acupuncture (AS Super 4 digital needle stimulator, Harmony Medical Co). They received 2 treatments per week for 4 weeks.
  Needle acupuncture (Traditional Acupuncture): This group received needle acupuncture at 3 pairs of sites. The needles were stimulated with low intensity, low frequency electric current using a constant-current electro-acupuncture device (AS Super 4 digital needle stimulator).
Period: Eligibility to Baseline Data Collection
Arm/Group | Controls | Mock Laser Acupuncture | Electro-Acupuncture
Started | 27 | 39 | 40
Completed | 26 | 39 | 40
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0
Period: Baseline Data Collection
Arm/Group | Controls | Mock Laser Acupuncture | Electro-Acupuncture
Started | 26 (No healthy volunteers were given any treatment as they were used for baseline comparison purposes.) | 39 | 40
Completed | 26 | 39 | 40
Not Completed | 0 | 0 | 0
Period: Intervention
Arm/Group | Controls | Mock Laser Acupuncture | Electro-Acupuncture
Started | 0 (Healthy controls were never intended to have interventions.) | 39 | 40
Completed | 0 | 38 | 38
Not Completed | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Baseline Analysis was done only for participants who completed trial.
Groups:
- Non-Traditional (Mock) Acupuncture: 39 fibromyalgia patients were randomized to non-traditional laser acupuncture (Vita Laser 650, Lhasa OMS).
  They received 2 treatments per week for 4 weeks. As consented, they were told, with IRB permission, that they were receiving laser acupuncture. This deception was essential to maintaining scientific integrity of the masking.
  Laser acupuncture (Non-traditional Acupuncture): For non-traditional acupuncture, a laser acupuncture device (Vita Laser 650, Lhasa OMS) was positioned over all of the same acupoints used in electro-acupuncture (EA), but was turned off during treatment sessions. There was no palpation prior to positioning these devices, and there was no physical contact between device and skin.
- Traditional Acupuncture: 40 fibromyalgia patients were randomized to receive electro-acupuncture (AS Super 4 digital needle stimulator, Harmony Medical Co). They received 2 treatments per week for 4 weeks.
  Needle acupuncture (Traditional Acupuncture): This group received needle acupuncture at 3 pairs of sites. The needles were stimulated with low intensity, low frequency electric current using a constant-current electro-acupuncture device (AS Super 4 digital needle stimulator).
- Total: Total of all reporting groups
Arm/Group | Controls | Non-Traditional (Mock) Acupuncture | Traditional Acupuncture | Total
Number analyzed (Participants) | 26 | 38 | 38 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.542881) | 41.5 (9.865814) | 44.5 (12.40337) | 43 (12.203111)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 38 | 38 | 102
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 7 | 2 | 1 | 10
  White | 19 | 31 | 35 | 85
  More than one race | 0 | 4 | 2 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 38 | 38 | 102

OUTCOME MEASURES:

1. Primary Outcome: Brain Neurocircuitry Underlying Chronic Pain (Percent of Time of a Somato-sensory Cortex Coactivation Pattern)
Description: Characterize the altered somatosensory-related neurocircuitry underlying chronic pain in FM, as shown by the difference in brain connectivity between healthy controls and FM patients as measured by FMRI (occurrence rate of co-activation pattern). For each arm, the coactivation pattern was assessed at rest and during a pressure pain stimulation.
  This is measured by the percent of scan time that an individual's brain displayed a particular coactivation pattern related to the somatosensory system.
Time Frame: At baseline
Population: Because this is at baseline (pre-treatment) all fibromyalgia patients are combined in a single analysis group. Some individuals' data was unable to be analyzed because of typical collection challenges (e.g. participant movement). Three participants were lost to follow-up. Four fibromyalgia patients were excluded due to: pain from shingles (N=1), starting Adderall treatment (N=1), inadequate treatments (N=1), and doubling pregabalin dosage (N=1), taking place during the study.
Measure: Mean (Standard Deviation); unit: percentage of scan time
Groups:
- Healthy Controls: Healthy pain free controls were recruited for comparison with fibromyalgia patients.
- Fibromyalgia Patients: All fibromyalgia patients measured at baseline (regardless of randomization).
Arm/Group | Healthy Controls | Fibromyalgia Patients
Number analyzed (Participants) | 19 | 63
percentage of scan time
  Sensorimotor co-activation pattern at rest | 0.1281 (0.05229) | 0.1190 (0.03835)
  Salience network co-activation pattern at rest | 0.1213 (0.05289) | 0.1345 (0.04560)
  Sensorimotor co-activation pattern at pressure pain | 0.1328 (0.05213) | 0.1362 (0.03972)
  Salience network co-activation pattern at pressure pain | 0.1121 (0.05065) | 0.1054 (0.04662)
Statistical Analysis 1: Comparison: Healthy Controls; Salience co-activation pattern at rest vs. with pressure pain; Test type: Superiority; p = 0.3330, t-test, 2 sided
Statistical Analysis 2: Comparison: Healthy Controls; This statistical analysis covers the sensorimotor co-activation pattern at rest vs. with pressure pain for Healthy controls; Test type: Superiority; p = 0.6474, t-test, 2 sided
Statistical Analysis 3: Comparison: Fibromyalgia Patients; Salience co-activation pattern at rest vs. with pressure pain; Test type: Superiority; p < 0.0001, t-test, 2 sided
Statistical Analysis 4: Comparison: Fibromyalgia Patients; This statistical analysis covers the sensorimotor co-activation pattern at rest vs. with pressure pain for Fibromyalgia patients; Test type: Superiority; p = 0.0004, t-test, 2 sided

2. Primary Outcome: Change in Brain Connectivity With Acupuncture Treatment
Description: Brain connectivity will be assessed at baseline and following either electro-acupuncture or mock laser acupuncture. Primary somatosensory cortex to insula connectivity. (Z-stat) A positive Z score reflects positive correlation in FMRI signal between different between brain areas. A negative Z score represents anti-correlation between in FMRI signal between brain regions. These scores reflect either positive connectivity or inhibitory connectivity. A mean of 0 represents no correlation or connectivity between regions.
Time Frame: Baseline and 4 weeks
Population: Of the 38 participants in each arm who completed the intervention, three participants from the traditional acupuncture arm and one from the mock laser acupuncture arm were excluded from analysis for reasons complicating treatment interpretation, (e.g. addition of a new pain symptom or addition of an external study treatment.) Three participants from the Traditional Acupuncture arm were excluded due to poor data quality at either the pre- or post-treatment scanning visit.
Measure: Mean (Standard Deviation); unit: Z - stat
Arm/Group | Mock Laser Acupuncture | Traditional Acupuncture
Number analyzed (Participants) | 37 | 32
Z - stat
  Baseline | 0.5492 (1.799) | -0.3013 (1.178)
  Post-treatment (4 weeks) | -0.08589 (1.182) | 1.125 (1.379)
Statistical Analysis 1: Comparison: Mock Laser Acupuncture; This is a comparison of Mock Laser Acupuncture pre-and post 4 weeks of treatment; Test type: Superiority; p = 0.0653, t-test, 2 sided
Statistical Analysis 2: Comparison: Traditional Acupuncture; This is a P value for the change in Traditional Acupuncture, pre and post 4 weeks of treatment; Test type: Superiority; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change in Brain Neurochemistry of Combined Glutamate and Glutamine (Glx) Within the Anterior Insular Cortex With Acupuncture Treatment
Description: Brain neurochemistry assessed at baseline and following either electro-acupuncture or mock laser acupuncture using proton magnetic resonance spectroscopy (1H-MRS) measures of combined glutamate and glutamine (Glx).
Time Frame: Baseline and 4 weeks
Population: Sixteen of the thirty-nine Non-Traditional Acupuncture treatment participants were excluded either for missing data or poor data quality while twenty-one of the forty Traditional Acupuncture treatment participants were excluded for missing data or poor data quality.
Measure: Mean (Standard Deviation); unit: AIU (arbitrary institutional units)
Groups:
- Non-Traditional (Mock) Acupuncture: 39 fibromyalgia (FM) patients were randomized to control mock laser acupuncture (Vita Laser 650, Lhasa OMS). They received 2 treatments per week for 4 weeks. As consented, they were told, with IRB permission, that they were receiving laser acupuncture. This deception was essential to maintaining scientific integrity of the masking.
  Laser acupuncture (Non-traditional Acupuncture): For non-traditional acupuncture, a laser acupuncture device (Vita Laser 650, Lhasa OMS) was positioned over all of the same acupoints used in electro-acupuncture (EA), but was turned off during treatment sessions. There was no palpation prior to positioning these devices, and there was no physical contact between device and skin.
Arm/Group | Non-Traditional (Mock) Acupuncture | Traditional Acupuncture
Number analyzed (Participants) | 23 | 19
AIU (arbitrary institutional units)
  Glx at baseline | 11.91 (1.005) | 12.11 (1.940)
  Glx at 4 weeks | 11.82 (1.042) | 11.88 (1.572)
Statistical Analysis 1: Comparison: Non-Traditional (Mock) Acupuncture; Glx statistical comparison; Test type: Superiority; p = 0.7399, t-test, 2 sided
Statistical Analysis 2: Comparison: Traditional Acupuncture; Glx statistical comparison; Test type: Superiority; p = 0.6226, t-test, 2 sided

4. Secondary Outcome: Change in Brain Neurochemistry of Gama-aminobutyric Acid (GABA) Within the Anterior Insular Cortex With Acupuncture Treatment
Description: Brain neurochemistry assessed at baseline and following either electro-acupuncture or mock laser acupuncture using proton magnetic resonance spectroscopy (1H-MRS) measures gama-aminobutyric acid (GABA).
Time Frame: Baseline and 4 weeks
Population: Fourteen of the thirty-nine Non-Traditional Acupuncture treatment participants were excluded either for missing data or poor data quality while twenty-two of the forty Traditional Acupuncture treatment participants were excluded for missing data or poor data quality.
Measure: Mean (Standard Deviation); unit: AIU (arbitrary institutional units)
Arm/Group | Non-Traditional (Mock) Acupuncture | Traditional Acupuncture
Number analyzed (Participants) | 25 | 18
AIU (arbitrary institutional units)
  GABA at baseline | 3.250 (0.9074) | 3.264 (0.4840)
  GABA at 4 weeks | 3.135 (0.6650) | 3.210 (0.8271)
Statistical Analysis 1: Comparison: Non-Traditional (Mock) Acupuncture; GABA statistical comparison; Test type: Superiority; p = 0.6344, t-test, 2 sided
Statistical Analysis 2: Comparison: Traditional Acupuncture; GABA statistical comparison; Test type: Superiority; p = 0.7985, t-test, 2 sided

5. Other Pre Specified Outcome: Predicting Response to Acupuncture Using Brain Neurochemistry
Description: Baseline neuroimaging outcomes of neurochemistry are used to predict subsequent response to electro-acupuncture and laser acupuncture.
Time Frame: Baseline
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Predicting Response to Acupuncture Using Brain Connectivity
Description: Baseline neuroimaging outcomes of connectivity are used to predict subsequent response to electroacupuncture and laser acupuncture.
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AE data for healthy volunteers was collected for visits 2 through 3, which were both within 3 days of each other, up to 4 days total. No further AE data was collected for the healthy volunteers. For fibromyalgia participants, in both treatment arms, AE data was collected at every visit, covering a period of at least 6 weeks and then for up to another 6 months.
Arm/Group | Controls | Non-Traditional (Mock) Acupuncture | Traditional Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/39 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/39 | 0/40
Other Adverse Events (participants affected / at risk) | 0/27 | 9/39 | 22/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Controls (N=27) | Non-Traditional (Mock) Acupuncture (N=39) | Traditional Acupuncture (N=40)
Nausea (Gastrointestinal disorders) | 0 | 4 | 3
Bruising (Vascular disorders) | 0 | 0 | 5
Pain Attack (Psychiatric disorders) | 0 | 0 | 2
Headache (Nervous system disorders) | 0 | 2 | 2
Migraine (Nervous system disorders) | 0 | 0 | 3
Ear Tenderness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Fibromyalgia Flare (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2
Leg Cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Muscle Burning (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT02064296/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT02064296/ICF_002.pdf